CLINICAL TRIAL: NCT00140088
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Confirm the Effectiveness and Safety of ALGRX 3268 in Pediatric Subjects.
Brief Title: Efficacy and Safety of ALGRX 3268 in Management of Needlestick Pain in Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3268-3-003-1
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Procedural Pain
Keywords: Needlestick pain; Venipuncture pain
MeSH Terms: conditions — Pain, Procedural

INTERVENTIONS:
Drug: ALGRX 3268

SUMMARY:
Minor needlestick procedures often cause significant pain and distress in pediatric patients yet interventions to reduce pain are used infrequently. ALGRX 3268 is a novel, single-use, prefilled, needle-free product that immediately delivers powdered lidocaine into the epidermis and provides local analgesia in 2-3 minutes. The purpose of this phase III, prospective, randomized, double-blind, placebo-controlled study is to investigate the efficacy, safety and tolerability of ALGRX 3268 versus placebo in pediatric patients aged 3 to 18 years undergoing venipuncture or peripheral venous canulation procedures. The trial will enroll approximate 504 evaluable subjects at centers located in the US.

DETAILED DESCRIPTION:
Management of pain due to minor procedures such as venipuncture or peripheral venous canulation still represents an unmet medical need, especially in pediatric setting. Current therapeutic products have a relatively delayed onset of analgesia of at least 10 minutes; moreover the most used products require application with at least 30-60 minutes prior to procedure. Development of ALGRX 3268 is aimed at addressing this unmet need in management of pain associated with needlestick procedures.

ALGRX 3268 (Previously known as PowderJect(R) Dermal Lidocaine) is used for local anesthesia to provide within 1-3 minutes painless needle or cathether insertion for blod drawing. ALGRX 3268 is a single-use disposable system, incorporating a drug cassette and glass cylinder into a single hand held device, with a button to actuate the system.

The purpose of this phase III, multicenter, prospective, randomized, double-blind, placebo-controlled study is to investigate the efficacy, safety and tolerability of ALGRX 3268 versus placebo in pediatric patients 3 to 18 years of age, who undergo venipuncture or peripheral venous canulation procedures. The trial will enroll approximate 504 evaluable subjects at centers located in the US.

Three age groups are enrolled: 3-7 years, 8-12 years, 13-18 years. Within each age group subjects are randomized to receive ALGRX 3268 0.5 mg/20 bar or pressure matched placebo. One to 3 minutes after administration of study treatment at the back of the hand or antecubital fosa, venipuncture is performed with a needle/Vacutainer, needle/syringe or "butterfly", at the discretion of the investigator.

Subjects 3-18 years are asked to assess pain on venipuncture using Wong-Baker FACES pain rating scale, anchored at 0 for "no hurt" and 5 for "hurts worst". Assessment of pain will be analyzed in each age group 3-7, 8-12, 13-18 and using Wong-Baker FACES pain rating scale.

Children in the middle (8-12) and older (13-18) age groups will also rate pain at the ACF and BOH using a 100 mm VAS anchored at 0 for "no pain" and at 100 for "extreme pain". Parent/legal guardian will evaluate child's level of pain on a 100 mm VAS anchored at 0, for "no pain", and at 100 for "extreme pain".

Safety ratings of skin are completed at 15 and 30 minutes following the procedure. AEs/SAEs will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children of either gender [M/F: 1:1] undergoing venipuncture or peripheral venous cannulation at the antecubital fossa or back of hand. Children must have sufficient cognitive skills to identify faces depicting extremes of pain on the Wong-Baker FACES Pain Rating Scale, (ages 3-12) and/or the extremes of pain on a 100 VAS (ages 8-18).
* Ages 3-7, 8-12, 13-18 years inclusive. Informed consent forms must have been approved by the appropriate IRB. Signed informed consent must have been granted by the parent/legal guardian and assent to participate should have been sought (either verbally or in writting) from each child.
* In females of childbearing potential who in the judgement of the investigator or designee were sexually active, a negative preganancy test must have been documented prior to enrollment. A negative urine preganancy test was required in all teenage girls over the age of 14 years. Surgically sterile females do not require a pregnancy test.

Exclusion Criteria:

* Previous history of allergic reactions to any local anesthetic. Any medical condition or instability that in the judgement of the investigator might have adversely impacted the conduct of the study and the collection of data.
* Subjects in whom the investigator determined that venipuncture could not be accomplished cleanly.
* Active local infection or other skin pathology on the dorsum of the hand. Subjects with tattos, surgical scars, ports, implantable devices or a skin condition that may have interfered with placement of study treatment or skin site assessments.
* Female subjects who were pregnant or lactating; females with a positive serum or urine pregnancy test; females of childbearing potential who were not using adequate contraception.
* Prior participation in an ALGRX 3268 study.
* Venipuncture at the proposed site within the prior 2 weeks (longer if bruising was apparent).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 504
Dates: Start 2004-12; Study Completion 2005-04

PRIMARY OUTCOMES:
Child's rating of pain on venipuncture following administration of the study treatment.

SECONDARY OUTCOMES:
Evaluation of pain due to venipuncture in each age group 3-7, 8-12 and 13-18.
Parent/legal guardian's rating of child's pain on an 100 VAS.

CONTACTS AND LOCATIONS:
Overall Officials: William Zempsky, MD, Principal Investigator — Connecticut Childrne's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Schmitz ML, Zempsky WT, Meyer JM. Safety and Efficacy of a Needle-free Powder Lidocaine Delivery System in Pediatric Patients Undergoing Venipuncture or Peripheral Venous Cannulation: Randomized Double-blind COMFORT-004 Trial. Clin Ther. 2015 Aug;37(8):1761-72. doi: 10.1016/j.clinthera.2015.05.515. Epub 2015 Jul 8. PMID 26164784
- [Derived] Zempsky WT, Bean-Lijewski J, Kauffman RE, Koh JL, Malviya SV, Rose JB, Richards PT, Gennevois DJ. Needle-free powder lidocaine delivery system provides rapid effective analgesia for venipuncture or cannulation pain in children: randomized, double-blind Comparison of Venipuncture and Venous Cannulation Pain After Fast-Onset Needle-Free Powder Lidocaine or Placebo Treatment trial. Pediatrics. 2008 May;121(5):979-87. doi: 10.1542/peds.2007-0814. PMID 18450903